CLINICAL TRIAL: NCT00001572
Title: Vaccination of Follicular Lymphomas With Tumor-Derived Immunoglobulin Idiotype
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970077; 97-C-0077; NCT00878410 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-02

CONDITIONS: B Cell Lymphoma; Follicular Lymphoma; Neoplasm
Keywords: B-Cell Lymphoma; BCL- 2 Positive Tumor; Immunization; Induction Chemotherapy; Lymphoma Vaccine; Follicular Lymphoma; Tumor-Derived Immunoglobulin Idiotype
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Neoplasms | interventions — saponin QA-21V1; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Id-KLH Vaccine
Drug: QS-21 (Stimulation-QS-21) Drug

SUMMARY:
Patients undergo chemotherapy until remission is obtained, or disease has been stable for two cycles of chemotherapy, or progressive disease develops.

Three to six months after completion of chemotherapy, patients who have achieved complete clinical remission or minimal disease status receive a series of 5 injections (given 1-2 months apart) of a vaccine consisting of 0.5 mg autologous tumor-derived immunoglobulin (Id) conjugated to KLH. The vaccine is administered with subcutaneous QS-21 as an immunological adjuvant....

DETAILED DESCRIPTION:
The idiotype of the immunoglobulin on a given B cell malignancy (Id) can serve as a clonal marker, and a previous pilot study in lymphoma patients has demonstrated that autologous Id protein can be formulated into an immunogenic, tumor specific antigen by conjugation to a carrier protein (KLH) and administration with an emulsion-based adjuvant.

The objectives of this study are: 1) to evaluate feasibility and toxicity of new vaccine formulations, and 2) to evaluate cellular and humoral immune responses against the unique idiotype of the patient's lymphoma.

The goal of this study is to treat patients with follicular lymphomas to complete remission or minimal residual disease with chemotherapy. Six to twelve months after completion of chemotherapy, in an effort to reduce the relapse rate (by eradicating microscopic disease resistant to chemotherapy), patients will receive one of two new formulations of an autologous Id vaccine.

ELIGIBILITY:
* INCLUSION CRITERIA:

Sample size: up to 30 patients.

Sex distribution: Male and female.

Age: Patients must be greater than or equal to 18 years old.

Patients must meet all of the following eligibility criteria:

Tissue diagnosis of: follicular small cleaved cell or follicular mixed lymphoma with surface IgM, IgA, or IgG phenotype with a monoclonal heavy and light chain. Pathology slides must be submitted to the NIH Pathology Department for review.

Stage III or IV lymphoma.

A single peripheral lymph node of at least 2x2 to 3x3 cm size and accessible for biopsy/harvest.

Karnofsky status greater than or equal to 70%.

Life expectancy of greater than 1 year.

Serum creatinine less than or equal to 1.5 mg/dl unless felt to be secondary to lymphoma.

Bilirubin less than or equal to 1.5 mg/dl unless felt to be secondary to lymphoma or Gilbert's disease. SGOT/SGPT less than or equal to 3.5 x upper limit of normal.

Ability to give informed consent. Ability to return to clinic for adequate follow-up for the period that the protocol requires.

There are no gender or racial / ethnic restrictions on patient selection. This protocol is open to all genders and racial / ethnic groups.

EXCLUSION CRITERIA:

The presence of any exclusion criteria (listed below) will prohibit entry onto study:

Prior total body irradiation.

Presence of antibodies to HIV or hepatitis B surface antigen or other active infectious process.

Pregnant or lactation. Fertile men and women must plan to use an effective contraception. A beta-HCG level will be obtained in women of child-bearing potential.

Patients with previous or concomitant malignancy, regardless of site, except curatively treated squamous or basal cell carcinoma of the skin, or effectively treated carcinoma in situ of the cervix.

Patient unwilling to give informed consent.

Failure to meet any of the eligibility criteria in Section 3.2.

Any medical or psychiatric condition that in the opinion of the protocol chairman would compromise the patient's ability to tolerate this treatment.

Patients with CNS lymphoma (current or previously treated) will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1997-01-30; Primary Completion 1999-07-31 (Actual); Study Completion 2010-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stevenson GT, Stevenson FK. Antibody to a molecularly-defined antigen confined to a tumour cell surface. Nature. 1975 Apr 24;254(5502):714-6. doi: 10.1038/254714a0. No abstract available. PMID 47617
- [Background] Sirisinha S, Eisen HN. Autoimmune-like antibodies to the ligand-binding sites of myeloma proteins. Proc Natl Acad Sci U S A. 1971 Dec;68(12):3130-5. doi: 10.1073/pnas.68.12.3130. PMID 4108872
- [Background] Kwak LW, Campbell MJ, Czerwinski DK, Hart S, Miller RA, Levy R. Induction of immune responses in patients with B-cell lymphoma against the surface-immunoglobulin idiotype expressed by their tumors. N Engl J Med. 1992 Oct 22;327(17):1209-15. doi: 10.1056/NEJM199210223271705. PMID 1406793